CLINICAL TRIAL: NCT03523871
Title: A Single-center Pilot Study of the Use of Hepatitis C Positive Donors for Hepatitis C Negative Lung Transplant Recipients With Post-transplant Treatment With Mavyret
Brief Title: A Study of the Use of Hepatitis C Positive Donors for Hepatitis C Negative Lung Transplant Recipients With Post-transplant Treatment With Mavyret
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-00091
Record Dates: First submitted 2018-04-11; First posted 2018-05-14 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir and pibrentasvir; pibrentasvir; glecaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Post Lung Transplant Patients (Experimental): The lung transplantation will be performed per standard of care techniques,and all post-transplant management of the transplanted organ, including immunosuppression, will be carried out per standard of care.
  Interventions: Drug: Mavyret

INTERVENTIONS:
Drug: Mavyret — Patients will be on 8 weeks of Mavyret
  Other Names: pibrentasvir; glecaprevir

SUMMARY:
Patients who are Hepatitis C Negative (HCV negative) and are on the waiting list for a lung transplant at NYULH who consent to participate in this study will receive a lung transplant from a deceased donor that is HCV positive. Patients will initiate treatment for HCV with the pan-genotypic agent, Mavyret, on the day of surgery and will complete the full 8-week treatment course. Patients will be monitored post-transplant for the development of viremia, and for the time course of clearance of viremia among those who develop viremia.

ELIGIBILITY:
Inclusion Criteria:

Recipient criteria:

* Listed for an isolated lung transplant at NYU Langone Health
* Between 18-70 years of age
* Able to travel to the NYU Langone Health for routine post-transplant visits and study visits for a minimum of 6 months after transplantation
* No active illicit substance abuse
* Weight at least 40kg
* Women of childbearing potential must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy (REMS) after transplant due to the increased risk of birth defects and/or miscarriage
* Both men and women must agree to use at least one barrier method after transplant to prevent any secretion exchange
* Able and willing to provide informed consent

Donor criteria:

* Detectable HCV RNA by nucleic acid test (NAT) or positive anti-HCV antibody
* Donor lung meets standard NYU Langone Health clinical criteria for procurement

Exclusion Criteria:

Recipient criteria:

* HIV positive
* HCV RNA positive or history of previously treated HCV
* Evidence of active hepatitis B infection or on active antiviral treatment for HBV
* Pregnant or nursing (lactating) women
* Use of strong CYP3A inducers
* Requires multi-organ transplant

Donor criteria:

* Confirmed HIV positive
* Confirmed HBV positive (positive hepatitis B surface antigen, and/or detectable Hepatitis B virus DNA)
* Known previously failed treatment for HCV
* Donor age >60 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-12 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Angel, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Post Lung Transplant Patients
Started | 20
Completed | 19
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Post Lung Transplant Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Incidences of Viremia After Receiving a Lung Transplant From a Donor Who Tests Positive for Hepatitis C
Description: Surveillance for the development of hepatitis C viremia post-transplant
Time Frame: 24 Months
Measure: Number; unit: incidences
Arm/Group | Post Lung Transplant Patients
Number analyzed (Participants) | 20
incidences | 16

2. Primary Outcome: Number of Patients With Sustained Virologic Response After Treatment
Description: HCV serologic testing to evaluate the presence of immunity to HCV or the evidence of prior infection with HCV.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Post Lung Transplant Patients
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Post Lung Transplant Patients
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post Lung Transplant Patients (N=20)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Post Lung Transplant Patients (N=20)
Increased shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Acute Renal Failure (Renal and urinary disorders) | 1
Right Hip Fracture (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT03523871/Prot_SAP_000.pdf